CLINICAL TRIAL: NCT06203860
Title: Cardiovascular Protection in Patients With Type 2 Diabetes and Established Heart or Vascular Disease - The Cardio-Metabolic Clinic
Brief Title: The Cardio-Metabolic Clinic
Acronym: ProtecT-2-D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ProtecT-2-D
Record Dates: First submitted 2023-12-10; First posted 2024-01-12 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus, Type 2; Cardiovascular Diseases
Keywords: Cardiovascular death; Heart attack; Stroke; Heart failure; Diabetic microvascular complications; Diabetic macrovascular complications
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Myocardial Infarction; Stroke; Heart Failure

STUDY DESIGN:
Intervention Model Description: Randomization in the ProtecT-2-D is carried out using the Randomization Module in the electronic Case Report Form (e-CRF) system, REDCap. To ensure concealed allocation the allocation table is created by a REDCap team member, who is independent of the ProtecT-2-D project staff.
  Participants will be randomized to either the Cardio-Metabolic Clinic or usual care in a ratio of 2:1
  1. Cardio-Metabolic Clinic
  2. Usual care
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Cardio-Metabolic Clinic (Active Comparator): Comprising specialized, multidisciplinary management of diabetes and cardiovascular disease in a Cardio-Metabolic Clinic.
  Interventions: Other: Cardio-Metabolic Clinic
- Usual Care (No Intervention): Involving collaboration between the general practitioner, and/or the endocrinology outpatient clinic, and/or cardiology outpatient clinic.

INTERVENTIONS:
Other: Cardio-Metabolic Clinic — The Cardio-Metabolic Clinic will adhere to a standardized evaluation and treatment program based on the latest treatment guidelines from the European Cardiovascular Society. The assessment will include the following points:
  * Lipid management
  * Blood pressure management
  * Antithrombotic therapy
  * Glycemic targets
  * Prevention of diabetes-related complications
  * Treatment of vascular disease affecting the lower extremities
  * Evaluation of cardioprotective drugs
  * Counseling on lifestyle factors, including diet, smoking, alcohol, and exercise
  * Guidance on vaccinations
  Arms: The Cardio-Metabolic Clinic

SUMMARY:
This study aims to investigate whether a Cardio-Metabolic Clinic can protect the cardiovascular health of patients with both diabetes and cardiovascular disease.

* At the Cardio-Metabolic Clinic, patients will receive a specialized and comprehensive care. This includes applying a systematic approach, considering their whole health based on the latest knowledge in the field, and administering aggressive treatment with heart protective medications.
* The ProtecT-2-D trial will compare the effects of care at the Cardio-Metabolic Clinic to usual care to see if there are any differences in cardiovascular illness and death.

DETAILED DESCRIPTION:
Background:

Despite improved treatment options, cardiovascular disease remains the leading cause of illness and death among patients with type 2 diabetes. It is crucial to recognize that managing diabetes involves more than just controlling blood sugar levels; preventing and treating cardiovascular disease is of significant importance. Lifestyle changes have been proven to have a substantial impact on cardiovascular health. Additionally, remarkable advancements in treatment options with cardiovascular protective effects have occurred over the past five years. Nevertheless, the traditional healthcare system primarily focuses on managing individual diseases, often leading to fragmented care for patients with type 2 diabetes. This fragmented approach often results in inadequate treatment, higher costs, and worse outcomes for cardiovascular disease. To address these challenges, our goal is to establish a Cardio-Metabolic Clinic that adopts a multidisciplinary approach to optimize diabetes management. The clinic will place special emphasis on implementing measures to protect the cardiovascular system and ensure comprehensive care for the patients. By bridging the gap between diabetes management and cardiovascular health, the aim is to enhance cardiovascular outcomes for patients with type 2 diabetes.

Organization in the Cardio-Metabolic Clinic:

The Cardio-Metabolic Clinic, structured on a cost-effective model, operates through a three-layered system centered on the patient. The innermost layer involves medical students or specialized cardio-metabolic nurses who maintain the daily contact with the patients. Patient medical history and baseline visit data are recorded in the Electronic Case-Report Form (Redcap). Upon randomization to the intervention arm, a decision-making algorithm in the Redcap-system is activated, ensuring that patients receive optimal and tailored medical treatment in accordance with the latest guidelines for diabetes management. The second layer includes a cardiologist who, in collaboration with the medical students or cardio-metabolic nurses, reviews the patients' risk profiles and algorithm-recommended treatments. If further counselling is needed for patient management, the third layer, consisting of an endocrinologist, a nephrologist and a hepatologist, will be consulted. This multidisciplinary collaboration ensures the most optimal diabetes management, especially in challenging cases.

Objectives:

The objective of the ProtecT-2-D trial is to investigate whether a comprehensive care in a Cardio-Metabolic Clinic are superior to standard treatment in reducing cardiovascular morbidity and mortality.

Hypothesis:

In patients with type 2 diabetes and cardiovascular disease, a systematic, specialized multidisciplinary approach in a Cardio-Metabolic Clinic, will result in better management of diabetes and reduced cardiovascular morbidity and mortality.

Methods:

The ProtecT-2-D study is a prospective, randomized, controlled trial conducted at the Cardiovascular Research Unit in Svendborg Hospital, Denmark. The study population consists of patients with type 2 diabetes and established cardiovascular disease, referred from general practices or seen in the outpatient clinic of Cardiology or Endocrinology at Svendborg Hospital. Sixteen hundred patients are anticipated to take part in the study. Patients are randomized in a 2:1 ratio to either receive comprehensive care at the Cardio-Metabolic Clinic or standard treatment. All patients are invited to undergo a health examination at baseline. Subsequently, patients enrolled in the Cardio-Metabolic Clinic will undergo a thorough multidisciplinary evaluation, including an optimization of lifestyle factors and medical treatment of cardiovascular risk factors based on current treatment guidelines.

After a duration of 3 years, all patients will be invited for a follow-up health examination. Furthermore, complications related to diabetes or cardiovascular disease will be assessed through registry and journal audits after 5 and 10 years.

Outcomes:

The primary outcome of the ProtecT-2-D trial is to investigate whether comprehensive care in a Cardio-Metabolic Clinic is superior to standard treatment. This will be assessed by the time to first occurrence of any of the endpoints in this composite: Death from cardiovascular causes, non-fatal myocardial infarction, non-fatal stroke, and hospitalization for HF.

Sample size estimation:

A reduction in the primary endpoint of 15 % is anticipated in patients assessed in the Cardio-Metabolic Clinic compared to standard treatment. With a power of 80% and an alpha value of 0.05, 1306 patients are needed, and a dropout rate of around 15-20% is anticipated; therefore, 1600 patients will have to be included in the study.

ELIGIBILITY:
Inclusion:

* >18 years
* Capable of giving written informed consent
* Established diagnosis of T2D
* Having established heart or vascular disease defined as either:
* Atherosclerotic disease defined as:

  1. Prior acute coronary syndrome (ACS).
  2. Chronic coronary syndrome defined as the combination of: Angina pectoris AND coronary atherosclerosis assessed with either Coronary CT angiography (CTA) or Myocardial-scintigraphy (MPI) or Coronary angiography (CAG) AND treatment with statins and/or acetylsalicylic acid.
  3. Stroke.
  4. Peripheral arterial disease (PAD) defined as: Claudication intermittence in combination with pathological ABI AND/OR vascular PAD surgery AND/OR ischemic amputation.
  5. Ischemic heart disease defined by one of the following criteria: a) Myocardial-scintigraphy: >10% reversibility OR b) Coronary CT angiography: Coronary Artery Calcium (CAC)-score >100.
* Heart failure (HF): HF with reduced ejection fraction (HFrEF), HF with Mildly reduced ejection fraction (HFmrEF), HF with preserved ejection fraction (HFpEF)
* Atrial fibrillation and/or flutter, including paroxysmal, persistent and chronic disease
* Valvular heart disease (which requires control in outpatient clinic of cardiology), such as aortic valve stenosis, mitral valve insufficiency, and patients with aortic dilatation
* Hypertension treated with at least three antihypertensive drugs

Exclusion:

* Life expectancy less than 5 years for any reason
* Type 1 Diabetes Mellitus
* Participation in another clinical trial with an investigational product or device that could interfere with the primary and/or secondary endpoints of this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2029-05-01 (Estimated); Study Completion 2034-05-01 (Estimated)

PRIMARY OUTCOMES:
Time to first occurrence of major adverse cardiovascular event (MACE), a composite endpoint consisting of: cardiovascular (CV) death, non-fatal myocardial infarction, non-fatal stroke, and hospitalisation for heart failure (HF). | From baseline to 5 years of follow-up
  Measured in days.

SECONDARY OUTCOMES:
Time to first occurrence of MACE, a composite endpoint consisting of: CV death, non-fatal myocardial infarction, non-fatal stroke, and hospitalisation for HF. | From baseline to 10 years of follow-up
  Measured in days.
Time to occurrence of the individual component CV death | From baseline to 5 and 10 years of follow-up
  Measured in days.
  Including: acute myocardial infarction, venous thromboembolic event, malignant arrhythmia, cardiogenic shock, fatal stroke and aorta dissection.
Time to occurrence of the individual component AMI. | From baseline to 5 and 10 years of follow-up
  Measured in days.
  Including: ST-elevation myocardium infarction and non-ST-elevation myocardium infarction
Time to occurrence of the individual component non-fatal stroke. | From baseline to 5 and 10 years of follow-up
  Measured in days.
  Including: Thromboembolic or undetermined
Time to first occurrence of a composite heart failure endpoint consisting of: de novo HF and HF hospitalisation. | From baseline to 5 and 10 years of follow-up
  Measured in days.
Number of overall symptom burden determined by summing the occurences of CV death, non-fatal myocardial infarction, non-fatal stroke, and hospitalisation for HF. | From baseline to 5 and 10 years of follow-up
  Measured in count of events.
Change in diabetic retinopathy stage based on eye examination (fundoscopy) | From baseline to 3 years of follow-up
  Measured in ratio to baseline.
Change in estimated Glomerular Filtration Rate (eGFR) | From baseline to 3 years of follow-up
  Measured in in ratio to baseline [mL/min/1.73 m^2]
  Creatinine-based.
Change in urinary albumin-to-creatinine ratio (UACR) | From baseline to 3 years of follow-up
  Measured in ratio to baseline.
Change in Chronic Kidney Disease (CKD) stage | From baseline to 3 years of follow-up
  Measured in ratio to baseline.
  Calculated by eGFR and albuminuria.
Time to first occurrence of a composite CKD endpoint consisting of a decline in eGFR [mL/min/1.73 m²] of more than 50%, onset of end-stage kidney disease (dialysis, eGFR<15, kidney transplantation) or death from renal or CV causes | From baseline to 3 years of follow-up
  Measured in count of events.
Change in fibrosis-4 (FIB-4) | From baseline to 3 years of follow-up
  Measured in ratio to baseline.
  FIB-4 is a biomarker assessing degree of liver fibrosis. Calculated using age, aspartate aminotransferase (ASAT), alanine aminotransferase (ALAT), and platelet count.
Change in degree of liver fibrosis in high-risk individuals assessed through a Fibro-scan | From baseline to 3 years of follow-up
  Measured in count of events.
Time to first occurrence of a composite macrovascular diabetic complications endpoint comprising new diagnosis of lower extremity arterial disease (LEAD), new/progression of foot ulcers, surgical procedures related to PAD, and coronary revascularisation | From baseline to 3 years of follow-up
  Measured in count of events.
  Surgical procedures in relation to PAD includes: percutaneous transluminal angioplasty, peripheral artery bypass, thrombectomy, thrombolysis, amputations.
  Coronary revascularisation includes: percutaneous coronary intervention (PCI), and/or coronary artery bypass graft.
Change in ankle-brachial pressure index (ABI). | From baseline to 3 years of follow-up
  Measured in ratio to baseline.
Change in protocol-driven medication | From baseline to 3 years of follow-up
  Measured in percentage (%).
  Protocol-driven medication includes:
  * Lipid lowering medication
  * Antihypertensive medication
  * Anti-thrombotic medication
  * Anti-diabetic medication
  * Nephro-protective medication
Change in symptoms as reported by patients using the Kansas City Cardiomyopathy Questionnaire (KCCQ) | From baseline to 3 years of follow-up
  Measured in score points (change in percentage [%])
Net cost analysis of implementing a Cardio-Metabolic Clinic | From baseline to 5 and 10 years of follow-up
  Measured in dollars [$].
  Cost of Cardio-Metabolic Clinic minus averted costs ( including averted admissions, medical treatment, and productivity).
Change in health outcomes measured by quality-adjusted life years (QALY) | From baseline to 5 and 10 years of follow-up
  Measured in score points (change in percentage [%])
Cost-effectiveness ratio of implementing a Cardio-Metabolic Clinic | From baseline to 5 and 10 years of follow-up
  Measured as: Net costs/change in health outcomes [$/QALY]

CONTACTS AND LOCATIONS:
Overall Officials: Soeren Auscher, M.D, Ph.D, Principal Investigator — Cardiovascular Research Unit. Odense University Hospital, Svendborg
Locations (1):
- Cardiovascular Research Unit, Odense University Hospital - Svendborg, Svendborg, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Overgaard KS, Mohamed RA, Andersen TR, Lambrechtsen J, Egstrup K, Auscher S. ProtecT-2-D trial protocol: cardiovascular protection in patients with type 2 diabetes and established heart and/or vascular disease at a cardio-metabolic clinic-a randomized controlled trial. Cardiovasc Diabetol. 2024 Jul 8;23(1):241. doi: 10.1186/s12933-024-02340-w. PMID 38978117